CLINICAL TRIAL: NCT01354067
Title: Effects of High-repetitive Single Limb Training on Exercise Capacity and Quality of Life in Patients With COPD Compared to a Control Group - A Prospective, Single Blind, Randomized Controlled Multicenter Trial
Brief Title: Single Limb Resistance Training in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Acronym: COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Responsible Party: Principal Investigator, Dr. Karin Wadell, Senior lecturer, Umeå University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LHM-2011-ANKW
Record Dates: First submitted 2011-05-11; First posted 2011-05-16 (Estimated); Last update posted 2012-06-21 (Estimated); Status verified 2012-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Pulmonary Disease, Chronic Obstructive; Lung Diseases, Obstructive; Single Limb; Elastic Resistance; Resistance Training; Minor Muscle Mass; Local muscle training
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases, Obstructive | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (Active Comparator): The control group will receive standardized patient education four times, once every two weeks, during the eight week intervention period.
  Interventions: Behavioral: Control group
- High-repetitive single limb training (Experimental): The experimental group will receive a high-repetitive single limb exercise regime, three times a week for two months. In addition, the exercise group will receive patient education at four occasions during the intervention period.
  Interventions: Behavioral: High-repetitive single limb training

INTERVENTIONS:
Behavioral: Control group — The control group receives standardized patient education four times, once every two weeks, during the eight week intervention period. Each session will last 60 minutes, consisting of information regarding anatomy, physiology, causes and mechanisms of COPD, drugs, nutrition, aids and energy saving procedures. The information is the same as for the intervention group, given at separate occasions.
  Arms: Control group
Behavioral: High-repetitive single limb training — The high-repetitive single limb exercise regime consists of three sessions per week during eight weeks of exercise training, giving a total number of 24 sessions at each location (Umeå and Huddinge University hospitals). The exercise sessions are supervised and conducted by a physical therapist using a group format, six to eight participants in each group. Each session will span for 60 minutes, duration of the major components are: 10 min warm-up followed by 40 minutes of single limb training and 10min cool-down. In addition this experimental group also receives four sessions of patient education once every two week.
  Arms: High-repetitive single limb training

SUMMARY:
The chronic airflow limitation in chronic obstructive pulmonary disease (COPD) patients resulting in increased dyspnea during physical activity restricts many COPD patients ability to perform exercises in general and whole-body exercises in particular. Single limb training performed as one-legged cycling has been shown effective in patients with COPD. This exercise regime results in less stress on the ventilatory system as training is executed using a simultaneously smaller muscle mass. However, the positive physiological effects of exercise training only occur in the involved muscle(s). To be of benefit for patients daily life, all relevant muscles should be included in exercise training. The aim of the current randomized controlled multicenter trial (RCT) is to determine the effects of high-repetitive single limb exercises (HRSLE) in combination with COPD specific patient education, compared to the COPD specific patient education alone in patients with moderate to very severe (stage II-IV) COPD.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a major cause of chronic morbidity and mortality in the world. It is one of our most common chronic diseases and up to 700.000 people is estimated to suffer from COPD in Sweden. Exercise intolerance is the key disabling factor in COPD, with decreased exercise capacity, leg fatigue and dyspnea among the most frequently reported symptoms.

Different training modalities have been evaluated to uncover the most effective way of training patients with COPD. Traditionally research has used whole-body, or major muscle mass training regimes when investigating the effect of both endurance and resistance in COPD patients. However recent research have demonstrated positive effects using training regimes involving a simultaneous smaller muscle mass compared to traditional exercise. The concept of using this regime is to put less stress on the ventilator system when exercising to minimize the effect of the chronic airflow limitation and to enhance the ability to be able to exercise for this group of patients compared to traditional training using major muscle mass exercise regimes. Although recent research have shown positive effects of single limb training using one-legged cycling, one major limitation is that only a small amount of important muscles for COPD patients are incorporated. Therefore, the aim of this study is to: (i) examine the effect of a single limb exercise regime on local muscle endurance, maximal strength, quality of life, dyspnea, walking capacity, self-efficacy, anxiety and depression, (ii) to examine if the physiological effects differ between man and women and (iii) to investigate if this exercise regime is feasible and safe to use for patients with COPD.

Patients diagnosed with moderate to very severe COPD according to GOLD criteria will be randomly assigned to constitute either an exercise or control group The exercise group will participate in a high-repetitive single limb exercise regime, consisting of upper and lower limb exercises with elastic resistance, compromised of three sessions per week over a period of 8 weeks. The exercise regime will be performed in group at Umeå University Hospital of Northern Sweden, and at Huddinge University Hospital, Sweden supervised by experienced physiotherapists. Both the exercise and control group will receive four sessions of standardized patient education during the 8 week intervention period. After completion of the study, patients in the control group will be offered participation in the single limb exercise regime.

The most important upper and lower extremity muscles for COPD patients are identified and exercises are designed specific to each of these. The exercise regime consists of 8 exercises, 4 upper extremity and 4 lower extremity exercises. Starting position and performance of the exercises are standardized and the resistance individually adjusted and progressed according to rated dyspnea and muscle fatigue.

Before and after the 8 week intervention period the following information will be collected. Effects on maximal strength, muscular endurance, dyspnea, self-efficacy, anxiety and depression. The relationship between changes in health related variables and changes in exercise capacity, sex related differences in training effects, feasibility of the program, strategies to determine adequate starting resistance and provide accurate resistance for each involved movement and the relationship between muscle fatigue and dyspnea in the different exercise tests will also be analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Adults 40 years and above.
2. Stable (no exacerbations within 4 weeks before start of baseline testing) moderate to very severe COPD, stage II-IV, according to GOLD criteria i.e. Forced expiratory volume in one second (FEV1)/ forced vital capacity (FVC) < 0.70, FEV1 < 80% predicted.
3. Ex-smoker.
4. Stable medical treatment (no changes < 4 weeks before start of baseline testing).
5. Living less than 60 km from training facility.

Exclusion Criteria:

1. Musculoskeletal, rheumatic, cardiac or neurological disorders that might affect the exercise performance in training and tests.
2. Previous lung surgery.
3. Acute exacerbations of COPD that require a change in pharmacological management within four weeks preceding the start of the intervention
4. Long-term oxygen treatment.
5. Participated in organized exercise training, > 2 times a week, within 6 months before start of intervention.
6. Body mass index (BMI) < 18 kg/m2.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2011-05; Primary Completion 2012-05 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Quality of life | Before single limb exercise regime and on completion (at 8 weeks)
  The Swedish Self-Administered Standardized version of the Chronic Respiratory Disease Questionnaire (CRQ-SAS) will be used as primary outcome measure to asses quality of life
Functional lower extremity muscular endurance | Before single limb exercise regime and on completion (at 8 weeks)
  To asses muscular endurance in the lower extremity the 6-minute walk test will be used as primary outcome measure.
Upper extremity muscular endurance | Before single limb exercise regime and on completion (at 8 weeks)
  The 6-minute ring and pegboard test will be used as primary outcome measure for upper extremity muscular endurance

SECONDARY OUTCOMES:
Isokinetic maximal muscle strength | Before single limb exercise regime and on completion (at 8 weeks)
  Maximal muscle strength in both upper and lower extremity will be evaluated with an isokinetic dynamometer
Upper extremity muscular endurance | Before single limb exercise regime and on completion (at 8 weeks)
  The Unsupported Upper Limb Exercise test will be used as secondary outcome measure for upper extremtiy muscular endurance
Isokinetic muscular endurance capacity | Before single limb exercise regime and on completion (at 8 weeks)
  Endurance capacity in both upper and lower extremity will be evaluated with an isokinetic dynamometer
Self-efficacy | Before single limb exercise regime and on completion (at 8 weeks)
  Self-efficacy will be evaluated with the exercise self-efficacy scale, and the self-efficacy for walking questionnaire
Anxiety and Depression | Before single limb exercise regime and on completion (at 8 weeks)
  Anxiety and Depression will be evaluated with the hospital anxiety and depression scale (HADs)
Relationship between muscle fatigue and dyspnea in the different exercise tests | Before single limb exercise regime and on completion (at 8 weeks)
  Muscle fatigue and dyspnea will be measured using the BORG CR10 scale during all exercise tests before the start of the study and on completion 8 weeks later. The relationship between ratings of muscle fatigue between tests, dyspnea between tests and the relationship between muscle fatigue rating and dyspnea rating between exercise tests will be investigated.
Develop a strategy to optimize resistance for each involved movement within an exercise regimen | Before single limb exercise regime and on completion (at 8 weeks)
  The exercises used within the intervention group is performed with elastic resistance. How much the elastic band is stretched for the different exercises is determined by a literature search investigation the strenght relationship between the muscles/movements used in the study. During the study each participant in the intervention group will rate muscle fatigue and dyspnea after each exercise during alla exercise sessions. These rating will be used to develop a strategy to optimize resistance for each involved movement within an exercise regimen
Develop a strategy to minimize attempts needed to determine a multiple repetition resistance using elastic bands | Before single limb exercise regime and on completion (at 8 weeks)
  55% of the isokinetic peak value obtained during baseline tests will be used to anticipate the 25RM load when using elastic resistance in an attempt to minimize the attempts needed to achieve 25RM.
Determine if this exercise regimen is feasible and safe in stage II-IV COPD patients | Before single limb exercise regime and on completion (at 8 weeks)
  Feasibility will be evaluated through number of participants attendance, adherence and number of participants developing any side effects or injuries during each training session. In addition, compliance to the different parts of the exercise regimen will be evaluated with a standardized questionnaire by both study participants and physiotherapists leading interventions.
Identify if there are any sex related differences in exercise training effects | Before single limb exercise regime and on completion (at 8 weeks)
  Statistical analyzes will be used to identify if there are any sex related differences in exercise training effects between male and female patients with COPD
Quality-of-life | Before single limb exercise regime and on completion (at 8 weeks)
  The clinical COPD questionnaire (CCQ) and the SF-36 scale will be used as secondary outcome measures for Quality-of-life
Exercise capacity | Before single limb exercise regime and on completion (at 8 weeks)
  A constant work rate test investigating the effects on endurance time, ventilatory response, perceived dyspnea and leg fatigue during submaximal cycle test.

CONTACTS AND LOCATIONS:
Overall Officials: Karin Wadell, Ph.D, Principal Investigator — Umeå University; Andre Nyberg, Msc, Study Chair — Umeå University; Britta Lindström, Ph.D, Study Chair — Umeå University
Locations (2):
- Sweden (2):
  - Huddinge University Hospital, Huddinge
  - Umeå University Hospital, Umeå

REFERENCES:
- [Derived] Nyberg A, Lindstrom B, Wadell K. Assessing the effect of high-repetitive single limb exercises (HRSLE) on exercise capacity and quality of life in patients with chronic obstructive pulmonary disease (COPD): study protocol for randomized controlled trial. Trials. 2012 Jul 23;13:114. doi: 10.1186/1745-6215-13-114. PMID 22823966